CLINICAL TRIAL: NCT00463619
Title: Follow-up Study With Retarded Release Phosphatidylcholine in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Other Study IDs: AVT123
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2010-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Retarded release phosphatidylcholine — 2g phosphatidylcholine, given QTD

SUMMARY:
Follow-Up Study with Retarded Release Phosphatidylcholine in Ulcerative Colitis

Objectives:

The objective of the study is to evaluate the follow up of patients treated with retarded release phosphatidylcholine in three controlled, randomized studies.

Main question is to investigate whether treatment with phosphatidylcholine could spare patients the intake of steroids and immunosuppressants without clinical deterioration.

Study population:

* Retarded release phosphatidylcholine in chronic-active ulcerative colitis.
* Retarded release phosphatidylcholine in steroid dependent ulcerative colitis.
* Dose finding study for retarded release phosphatidylcholine

Outcome parameters:

Definition of remission:

1. SCCAI <2,5
2. Likert scale: grade 1 or 2
3. subjective impression of remission: yes/no
4. no blood in stool

Definition of relapse:

1. subjective impression: yes/no
2. SCCAI ≥ 5
3. blood in stool

Definition of low clinical activity: SCCAI < 5

Primary endpoint:

sparing effect of steroids and/or immunosuppressants by rPC in chronic active UC.

Secondary endpoints

1. maintenance of continuous remission
2. improvement of disease activity: a. clinical activity (SCCAI) b.life quality (SIBDQ-D) c.Likert Score
3. relapse rate: a. time to first relapse b. clinical activity during relapses c. number of relapses in relation to length of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients from previous studies with retarded release phosphatidylcholine

Exclusion Criteria:

* patients with less then 6 weeks follow-up after end of initial study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from previous studies with retarded release phosphatidylcholine
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2000-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Karner, MD, Study Chair — University Heidelberg - Gastroenterology; Verena Schmieg, Cand. med., Principal Investigator — Heidelberg University
Locations (1):
- University Heidelberg - Dep. Gastroenterology, Heidelberg, Germany